### NCT04015167

# T2 Alpha Tibia Statistical Analysis Plan (SAP)

CLINICAL INVESTIGATION

TITLE:

A Post-Market Clinical Evaluation of the Treatment of Tibia

Fractures with the T2 Alpha Tibia Nailing System

**DEVICE NAME:** T2 Alpha Tibia Nailing System

STATISTICAL ANALYSIS PLAN

(SAP) VERSION:

3

**CLINICAL INVESTIGATION** 

PLAN (CIP) VERSION:

3

**INDICATIONS:** This clinical investigation will adhere to the indications and

contraindications for the T2 Alpha Tibia Nailing System as are

detailed in the device's Instructions For Use.

CLINICAL INVESTIGATION

**DESIGN:** 

• Post-Market,

• Multicenter,

• Prospective,

• Non-Randomized

CONFIDENTIALITY STATEMENT:

This Statistical Analysis Plan contains confidential information and its' use is limited to investigational staff intending to conduct the clinical investigation, Institutional Review Boards

(IRBs)/Ethics Committees (ECs) and any others charged with

reviewing the clinical investigation.

**DATE:** July 23<sup>rd</sup> 2021

# **Approval Page**

| APPROVERS | | | | |
|---|---|---|---|---|
| Role | Name | Signature | | Date |
| Author | Sascha Lorenzen | Sascha Lorenzen | Electronicall<br>y signed by:<br>Sascha<br>Lorenzen<br>Reason: I<br>am signing<br>as the<br>Author of<br>this<br>document<br>Date: Jul 23,<br>2021 12:15<br>GMT+2 | 23-Jul-2021 |
| Statistician | Claudia Beimel | Bernel | Electronical ly signed by: Claudia Beimel Reason: I approve this document Date: Jul 23, 2021 13:19 GMT+2 | 23-Jul-2021 |
| Clinical Research<br>Head (CRH) | Rebecca Gibson | Rebecca Jibson | Electronical ly signed by: Rebecca Gibson Reason: I approve this document Date: Jul 23, 2021 12:35 EDT | 23-Jul-2021 |
| Clinical<br>Investigation<br>Manager (CIM) | Susanne Hoefer | Susanne Höfer | Electronicall<br>y signed by:<br>Susanne<br>Höfer<br>Reason: I<br>approve this<br>document<br>Date: Jul<br>23, 2021<br>12:36<br>GMT+2 | 23-Jul-2021 |

# **Table of Contents**

| 1. | Admini | strative Information | 5 |
|----|---------|----------------------------------------------------|----|
| | 1.1. | LIST OF ABBREVIATIONS | 5 |
| | 1.2. | STATISTICAL ANALYSIS PLAN REVISION HISTORY | 5 |
| | 1.3. | ROLES AND RESPONSIBILITIES | 6 |
| 2. | Introdu | ıction | 6 |
| | 2.1. | BACKGROUND AND RATIONALE | 6 |
| | 2.2. | CLINICAL INVESTIGATION DESIGN | 6 |
| 3. | Researc | ch Goals | 6 |
| | 3.1. | FRAMEWORK | 6 |
| | 3.2. | SAMPLE SIZE | 9 |
| 4. | Method | ls | 12 |
| •• | 4.1. | RANDOMIZATION | |
| | 4.2. | STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE | 12 |
| | 4.3. | TIMING OF FINAL ANALYSES | |
| | 4.4. | TIMING OF OUTCOME ASSESSMENT | 12 |
| | 4.5. | STATISTICAL SOFTWARE | 13 |
| | 4.6. | MISSING DATA | 13 |
| | 4.7. | CONFIDENCE INTERVALS AND P-VALUES | 13 |
| | 4.8. | UNITS | 14 |
| | 4.9. | CALCULATIONS AND TRANSFORMATIONS | 14 |
| | 4.10. | ASSUMTIONS | 14 |
| 5. | Popula | tion and Progress | 14 |
| | 5.1. | ANALYSIS POPULATION | 14 |
| | 5.2. | ELIGIBILITY | 15 |
| | 5.3. | WITHDRAWAL / FOLLOW-UP | 15 |
| | 5.4. | ADHERENCE AND CIP DEVIATIONS | 15 |
| 6. | Analysi | is | 16 |
| | 6.1. | HARMS AND SAFETY | 16 |
| | 6.2. | BASELINE CHARACTERISTICS | 17 |
| | 6.3. | INTRA-OPERATIVE CHARACTERISTICS | 23 |
| | 6.4. | EARLY POST-OPERATIVE CHARACTERISTICS | 24 |
| | 6.5. | POST-OPERATIVE CHARACTERISTICS | 24 |
| | 6.6. | ANALYSIS OF CI ENDPOINTS | 29 |

| | 6.7. | ADDITIONAL ANALYSIS | 30 |
|---|---|---|---|
| | | <ul> <li>6.7.1. SF-36 Total Physical Score Comparison.</li> <li>6.7.2. Weight-bearing status.</li> <li>6.7.3. External Support.</li> <li>6.7.4. Mortality.</li> <li>6.7.5. Revision Surgery.</li> <li>6.7.6. SF-36 Total Physical Score – Within subject changes by visit.</li> </ul> | 31<br>32<br>34 |
| 7. | Table T | Геmplates (Tables, Figures, Listings - TFL) | 37 |
| | 7.1. | FREQUENCIES | 37 |
| | 7.2. | DESCRIPTIVE STATISTICS | 37 |
| | 7.3. | LISTINGS | 38 |
| 8. | Referei | nces | 39 |

# 1. Administrative Information

### 1.1. LIST OF ABBREVIATIONS

| <u>Acronym</u> | <b>Definition</b> |
|---|---|
| ADE | Adverse Device Event |
| AE | Adverse Event |
| CI | Confidence Interval |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| eCRF | Electronic Case Report Form |
| EC | Ethics Committee |
| EDC | Electronic Data Capture |
| EU MDR | European Medical Device Regulation |
| FR | Final Report |
| ICF | Informed Consent Form |
| ICH-GCP | International Conference of Harmonisation Good Clinical Practice |
| IFU | Instructions for Use |
| ITT | Intent-to-Treat |
| Intra-Op | Intra-Operative |
| IR | Interim/Annual Report |
| IRB | Institutional Review Board |
| LTFU | Lost to Follow-Up |
| MCS | SF-36 Mental Component Summary |
| PCS | SF-36 Physical Component Summary |
| PP | Per Protocol |
| Pre-Op | Pre-Operative |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SF-36v2 | 36-Item Short Form Health Survey |
| UADE | Unanticipated Adverse Device Effect |

### 1.2. STATISTICAL ANALYSIS PLAN REVISION HISTORY

| Version | Effective Date | Description | Reason |
|---|---|---|---|
| 1 | 25MAR2020 | Initial Version | |
| 2 | 24JUL2020 | Adjustment chapter 4.4<br>Timing of Outcome<br>Assessment | CIP changes, merge of<br>Pre-Operative and<br>Operative/ Discharge<br>visit. |
| 3 | 23JUL2021 | Distinction<br>interim/final Analysis<br>Amendment Table<br>Templates section 7 | Revision DQI 20-048,<br>CIP V3 |

| CIP changes: chapter 2.2 |
|--------------------------|

#### 1.3. ROLES AND RESPONSIBILITIES

| Role | Contributor | Affiliation |
|--------------------------------------|-----------------|-------------|
| Author | Sascha Lorenzen | Stryker |
| (Senior) Statistician | Claudia Beimel | Stryker |
| Clinical Research Head (CRH) | Rebecca Gibson | Stryker |
| Clinical Investigation Manager (CIM) | Susanne Hoefer | Stryker |

### 2. Introduction

#### 2.1. BACKGROUND AND RATIONALE

The T2 Tibia Nailing System represents the latest and most comprehensive development of the original intramedullary principles presented by Professor Gerhard Kuentscher in 1940. As an addition to the T2 Nailing System, Stryker has created a new generation tibial implant that offers an efficient treatment option for multiple indications. The T2 Alpha Tibia Nail includes new locking options and the ability to utilize the advanced locking screw which creates an axial and angular stable construct. New instrumentation offers a combination of innovation, simplicity and efficiency that is designed to suit the various needs of surgeons and OR staff.

The T2 Alpha Tibia Nailing System is fully integrated into the T2 Alpha Platform. The system includes two approaches: infrapatellar approach and suprapatellar approach and allows for multiple locking configurations for stable fixation. This clinical investigation will evaluate the safety and efficacy/performance of the T2 Alpha Tibia Nailing System.

### 2.2. CLINICAL INVESTIGATION DESIGN

This investigation is a prospective, multicenter clinical investigation. It is anticipated that a total of 80 subjects will be enrolled at up to 5 sites. Enrollment is estimated to commence in Q4 of 2018. Neither subjects nor investigators are blinded to treatment and the clinical investigation includes a historical control which will be compared to the T2 Alpha Tibia Nailing System.

The enrollment period is expected to occur over 32 months. Total duration of enrollment, 12 month follow-up and analysis is expected to take 47 months. The clinical investigation has been designed to follow the surgeon's standard of care for tibia fractured subjects, in addition to a 12 month follow-up visit.

### 3. Research Goals

### 3.1. FRAMEWORK

All quantitative variables, including those based on calculations (secondary elements), will be analyzed with a case summary evaluation before the detailed characteristics and parameter can be evaluated. A case summary contains a listing of the number of valid cases/values, missing cases/values (if any) and total cases/values in the specific analysis. In general, as central position parameter for quantitative

variables the mean and median will be analyzed. As variation parameter the standard deviation, 95% confidence interval of the mean, interquartile range and maximum and minimum will be calculated. All quantitative variables will be assessed for normality used the Shapiro-Wilk test. For optional visualization of quantitative variables, box-and-whisker plots will be used. Additional analyses like skewness and kurtosis measures of standard errors are also optional.

All qualitative variables, including those based on summaries (secondary elements), will be analyzed listing the proportions, frequencies, column and row totals and missing proportion (if any).

### 3.1.1. Primary Analysis / Endpoint

This analysis is only part of the final report. The primary endpoint analysis will only be executed once at the end of the clinical investigation and will not be part of any interim or annual reports or presentations given in front of the final report.

The 12 months post-operative results for subjects implanted with the T2 Alpha Tibia Nailing System will be compared to Sanders et al: Semiextended intramedullary nailing of the tibia using a suprapatellar approach: radiographic results and clinical outcomes at a minimum of 12 months follow-up. J Orthop Trauma, 2014; Sun et al: The outcome comparison of the suprapatellar approach and infrapatellar approach for tibia intramedullary nailing. Int Orthop, 2016; and Chan et al: Suprapatellar Versus Infrapatellar Tibial Nail Insertion: A Prospective Randomized Control Pilot Study. J Orthop Trauma, 2016". Specifically, the SF-36 score results reported by Wang, et al. (2017), Sanders, et al. (2014), Sun, et al. (2016) and Chan, et al. (2016) will serve as the control groups for the T2 Alpha Tibia group.

Higher SF-36 PCS and MCS score results are linked to better subject results and vice versa.

The clinical investigation endpoint is non-inferiority to the control, meaning the clinical investigation result should be equal or better than the control. In this clinical investigation, an equal or better SF-36 score result means equal or greater ( $\geq$ ). As only results from samples will be captured, results are mostly estimates of the true population parameter. These estimates vary by a certain area, where it is expected that the true population parameter falls within. Based on this, it is required to specify a lower limit for the acceptable difference or zone of indifference, denoted as  $-\theta$ .

Hypotheses were developed to allow for a comparison of the 12 months post-operative SF-36 PCS to evaluate effectiveness / performance. The 12 months post-operative SF-36 PCS is the primary endpoint of this clinical investigation. Hypothesis tests will be one-sided with a significance level  $\alpha$  of 5%.

| Hypothesis | Equations | Interpretation |
|---|---|---|
| Null (H <sub>0</sub> ) | A – B < -θ T2 Alpha Tibia (A) – Control (B, pooled benchmark results) < -θ | Central tendency of A is inferior to the central tendency of B. |
| Alternative (H <sub>1</sub> ) | $A - B ≥ -\theta$ T2 Alpha Tibia (A)- Control (B, pooled benchmark results) ≥ -θ | Central tendency of A is non-inferior to the central tendency of B. |



To test non-inferiority, the 12 months mean SF-36 PCS result of the T2 Alpha Tibia group will be compared to the mean estimate of the control group, 43.48 points.

To be able to identify an acceptable difference or zone of indifference (-θ), the lower 90% confidence interval (CI) of the SF-36 PCS result at 12 months post-operative in the control group (Sanders, et al.; Sun, et al.; Chan, et al.) was used as lower limit (lower 90% CI of control is 39.25 points). The maximum acceptable difference in the negative direction is 4.23 points.

Based on the underlying distribution of the data and the result of the normality assessment, either the parametric one-sample t-test or the non-parametric one-sample sign test will be used to compare the 12 months post-operative SF-36 PCS result of the T2 Alpha Tibia group against the value of 39.25 points (mean of control -  $\theta$  or 43.48 – 4.23 = 39.25 points).

#### 3.1.2. Secondary Analyses

For efficacy/performance, bone consolidation will be assessed by 12 months as measured by Investigator assessment. For Safety, the incidence of device-related adverse events/incidents by 12 months will be monitored through collection and analyses. Both analyses will be part of the final report.

Furthermore, device related adverse events/incidents and the time to (earliest) Device Related Adverse Events/incidents will be analyzed as well. Considered variables, the level of measurement and the planned analysis steps are listed in detail in the SAP.

### 3.1.3. Additional Analyses

Additional Analyses are outlined in the subsequent sections. Analysis details (variables, level of measurement, planned steps) are listed in-depth in the SAP.

### Weight-bearing status

The weight bearing status will be evaluated and analyzed at the pre-operative visit and at 3 months, 6 months and 12 months. The within subject changes from visit to visit will be analyzed in addition. This analysis will be part of the final report.

### External Support

The status of the subject using external support will be evaluated at the pre-operative visit and at 3 months, 6 months and 12 months. The within subject changes from visit to visit will be analyzed in addition. This analysis will be part of the final report.

### Mortality

For analysis of the time to death or mortality, the Kaplan-Meier method will be used. The times between the date of surgery and the date of the 12 months assessment will be used together with the times between date of surgery and the date of death. This analysis will be part of the final report.

### Reoperation

For analysis of the time to the reoperation, the Kaplan-Meier method will be used. The times between the date of surgery and the date of the 12 months assessment will be used together with the times between date of surgery and the date of reoperation (earliest reoperation in case that one subject experienced more than one reoperation). This analysis will be part of the final report.

### SF-36 Total Physical Score – Within subject changes by visit

The within subject score changes of the SF-36 Total Score from visit to visit will be analyzed to help identify the changes on the subject level. This analysis will be part of the final report.

### 3.2. SAMPLE SIZE

The 12 months post-operative results for subjects implanted with the T2 Alpha Tibia Nail will be compared to a historical group and results reported by Wang, et al. (2017); Sanders, et al. (2014); Sun, et al. (2016); and Chan, et al. (2016) will serve as the control group for the T2 Alpha Tibia Nail subjects.

Hypotheses were developed to allow for a comparison of 12 months post-operative SF-36 Physical Component Summary (PCS) results and 12 months effectiveness/performance between these two populations.

| Benchmark and Objectives for Planned Research | |
|---|---|
| Endpoint | Non-inferiority related to the SF-36 Physical Component Summary (PCS) for subjects undergoing infrapatellar (IP) and/or suprapatellar (SP) tibia nailing at 12 months post-operative compared to the pooled literature control. |
| Estimated drop-<br>out rate | 20% Source: "Stannard et al: Functional Outcome Following Intramedullary Nailing of the Tibia. A Prospective Randomized Comparison of Piriformis Fossa and Greater Trochanteric Entry Portals JBJS 2011" Stannard et al. reported a lost to follow up rate of 19.6% (11/56). Note: The source of Stannard et al. was used for T2 Alpha Tibia as well as it represents a worst-case drop-out rate. |

### Results as reported by Benchmark

Non-inferiority related to the SF-36 Physical Component Summary (PCS) for subjects undergoing infrapatellar (IP) or suprapatellar (SP) tibia nailing at 12 months post-operative.

The results from the sources Chan et al, Sanders et al., and Sun et al. were pooled to determine overall two-sided 90% confidence intervals of the mean SF-36 PCS (physical) and mean SF-36 MCS (mental) scores.

Note: The results reported by Wang et al. seemed to be based on a different calculation method for the determination of the SF-36 scores and it was not possible to evaluate, what exactly was done by the authors. The score values reported by Wang et al. are much higher compared to what was normally reported in the literature and what was defined in country specific weights and coefficients. Wang et al. reported median

score values whereas the other authors reported means. As summary score results usually tend to deviate from normality, means and medians might differ significantly. Therefore, the results reported by Wang et al. were not included into the pooled analysis.

| Source | Subgroup | Mean SF36-<br>PCS | Mean SF36-<br>MCS | Pooling |
|----------------|----------|-------------------|-------------------|----------|
| Chan et al. | IP | 38.00 | 47.00 | included |
| Chan et al. | SP | 46.00 | 47.00 | included |
| Sanders et al. | SP | 40.80 | 46.00 | included |
| Sun et.al. | SP | 49.41 | 44.71 | included |
| Sun et.al. | IP | 43.21 | 43.81 | included |
| Wang et.al. | | 79.10 | 77.00 | excluded |

Summary of explorative analysis is listed below:

#### Descriptives

| | | | Statistic | Std. Error |
|---|---|---|---|---|
| SF-36 PCS Physical at 12 | Mean | | 43,4840 | 1,98495 |
| months post-op | 90% Confidence Interval | Lower Bound | 39,2524 | |
| | for Mean | Upper Bound | 47,7156 | |
| | Median | | 43,2100 | |
| | Std. Deviation | | 4,43849 | |
| | Minimum | | 38,00 | |
| | Maximum | | 49,41 | |
| | Range | | 11,41 | |
| | Interquartile Range | | 8,31 | |
| SF-36 PCS Mental at 12 | Mean | | 45,7040 | ,63333 |
| months post-op | 90% Confidence Interval | Lower Bound | 44,3538 | |
| | for Mean | Upper Bound | 47,0542 | |
| | Median | | 46,0000 | |
| | Std. Deviation | | 1,41617 | |
| | Minimum | | 43,81 | |
| | Maximum | | 47,00 | |
| | Range | | 3,19 | |
| | Interquartile Range | : | 2,74 | |

As the mean physical score (PCS) was slightly lower, it was used for the sample size calculation.

For the clinical investigation the one-sided 95% confidence interval will be applied.

| Acceptance Criteria for Sample Size Calculation | | |
|---|---|---|
| Significance Level (α) | 0.05 (5%) | |
| Power (1-β) | 0.80 (80%) | |
| Confidence Interval (CI) | 0.95 (95%) | |
| Tails | 1 | |
| Path | Non-inferiority T2 Alpha Tibia (A) ≥ Benchmark (B, pooled benchmark results) | |
| Hymothogog Doin | Null (H <sub>0</sub> ) | $A - B < -\theta$ |
| Hypotheses Pair | Alternative (H <sub>1</sub> ) | $A-B \ge -\theta$ |
| Benchmark Timepoint | 12 months post-operative | |
| Benchmark Mean | 43.48 points SF-36 PCS at 12 months (IP and SP together) | |
| | No standard deviation results were given by Chan et al., Sanders et al. nor Wang et al. | |
| Benchmark Std. Dev. | • Only Sun et al. reported standard deviations at 12 months postoperative for SF-36 PCS of 6.27 for the SP and of 6.52 for the IP subgroup | |
| | As a worst-case, the double standard deviation reported by Sun et al. was usefor the sample size calculation $(2 * 6.52 = 13.04 \text{ points})$ | |
| Benchmark 90% CI of Mean | <b>Lower 90% CI: 39.25</b> (two-sided 90% CI equals a one-sided 95% CI) | |

| | Upper 90% CI: 47.72 |
|---------------|----------------------------------|
| Margin (-θ) | Lower 90% CI of Benchmark: 39.25 |
| Software Used | IBM SPSS Sample Power V3.0 |

### **IBM SPSS Sample Power Output**

One goal of the proposed clinical investigation is to test the null hypothesis that the population mean is 39.25. The criterion for significance (alpha) has been set at 0.050. The test is 1-tailed, which means that only an effect in the expected direction will be interpreted.

With the proposed sample size of 61 subjects, the clinical investigation will have power of 80.0% to yield a statistically significant result.

This computation assumes that the population from which the sample will be drawn has a mean of 43.48 with a standard deviation of 13.04. The observed value will be tested against a theoretical value (constant) of 39.25.

This effect was selected as the smallest effect that would be important to detect, in the sense that any smaller effect would not be of clinical or substantive significance.

A second goal of this clinical investigation is to estimate the mean in the population. On average, a clinical investigation of this design would enable us to report the mean with a precision (95.0% confidence level) of plus/minus 2.77 points.

The precision estimated here is the median precision. Precision will vary as a function of the observed standard deviation (as well as sample size), and in any single clinical investigation will be narrower or wider than this estimate.

### IBM SPSS Sample Power Output – Screenshot



Estimated drop-out rate is 20% which leads to the requirement of enrolling additional 13 subjects into the clinical investigation.

| Sample Size | Overall number of subjects to be enrolled: 74 subjects (rounded up to 80 subjects) |
|---|---|

Table 3.2: Sample Size Justification

### 4. Methods

### 4.1. RANDOMIZATION

No specific methods for assigning subjects will be used for this clinical investigation. A consecutive series of subjects at each site meeting all the eligibility criteria will be enrolled in this clinical investigation.

### 4.2. STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE

Interim analyses will be performed on a yearly basis. The progress of the clinical investigation will be reported together with the interim results on the variable level according to the analysis plan.

As the primary endpoint analysis will only be conducted at the end of the clinical investigation, no adjustment of the significance level will be required.

There will be no stopping rules specified for this clinical investigation.

### 4.3. TIMING OF FINAL ANALYSES

The full final report with complete analyses, progress and conduct reporting will be created at the end of this clinical investigation.

### 4.4. TIMING OF OUTCOME ASSESSMENT

Subjects in this clinical investigation will be evaluated at Operative/Discharge, and at 3 Months, 6 Months and 12 Months after the index procedure. The follow-up evaluations will include assessment of device-related adverse events/incidents, evaluation per SF-36 PCS and MCS scores as well as clinical assessment of bone consolidation. Investigators should consider weight-bearing, pain and imaging when assessing bone consolidation. See the section below for visit windows and a list of assessments to be performed at each visit, given by the CIP.

| Assessment | Operative/<br>Discharge | 3 Months <sup>a, b</sup> (+/-2 weeks) | 6 Months <sup>a, b</sup> (+/-3 weeks) | 12 Months <sup>b</sup> (+/-4 weeks) |
|---|---|---|---|---|
| Informed Consent | X <sup>c</sup> | | | |
| Demographics & Medical History | X | | | |
| Inclusion/Exclusion | X | | | |
| Primary Diagnosis | X | | | |
| Surgical Procedure | X | | | |
| Clinical Assessment of Bone<br>Consolidation d, e | | X | X | X |
| SF-36v2 (PCS & MCS) | X f | X | X g | X g |
| Subject Disposition h | | X | X | X |

Device-Related Adverse Events/Incidents & Reoperations will be collected throughout the course of the Clinical Investigation.

- a. Follow-up visit schedule to reflect Institutions' Standard of Care practices
- b. If the subject missed a visit and outside of visit window, every effort should be made to collect data instead of noting visit as missed. Visit windows are calculated from the index event, and not from the previous visit.
- c. Informed consent must be obtained prior to enrollment in the study (i.e., prior to performance of any study-related activities).
- d. Once bone consolidation is observed, assessment no longer needs to be conducted at the additional follow-up visits.
- e. Investigators should consider weight-bearing, pain and imaging when assessing bone consolidation.
- f. SF-36v2 evaluation must be collected post-informed consent. This can be collected post-fracture and prior to surgery or immediately post-surgery.
- g. If bone consolidation is previously observed at the previous follow-up visit, evaluation is to be collected via phone.
- h. Subject Disposition assessment would occur at any time point for subject withdrawal prior to the completion of the clinical investigation.

Table 4.4: Assessments and Clinical Investigation Elements

In addition, the "Operative/Discharge" visit also includes Pre-operative data, which can also be recorded post-operatively, as defined in the CIP. Pre-operative- and operative data is aggregated as "Initial Assessment" in EDC frontend, but separately listed in EDC data exports for analysis. The pre-operative data is captured at "Primary Diagnoses" assessment, operative data at "Surgical Procedure" assessment. The SAP relates to the separate designation pre-operative- and operative assessment, as given by EDC export.

#### 4.5. STATISTICAL SOFTWARE

Statistical Analysis will be performed using IBM SPSS, IBM SPSS Sample Power as well as established standard software packages (e.g. MS Excel).

### 4.6. MISSING DATA

The intent is to collect as complete a dataset as possible. Nevertheless, in some situations missing data cannot be avoided. The reports and tables therefore will show the number and percentage of missing cases for each analyzed variable in relation to the enrolled cases for each post-operative assessment.

Missing data will be reported for each variable or calculation (if any) and overall totals will be reported including the proportion of missing data (if any).

### 4.7. CONFIDENCE INTERVALS AND P-VALUES

The following acceptance / rejection criteria were used for this clinical investigation:

| Parameter | Acceptance / rejection criteria |
|---------------------------------|---------------------------------|
| Confidence level (1-α) | 0.95 (95%) |
| Significance level (α) | 0.05 (5%) |
| Power (1-β) | 0.80 (80%) |
| Beta-level (β) | 0.20 (20%) |
| Confidence interval of mean | 95% |
| p-value indicating significance | ≤ 0.05 |

Table 4.7: Acceptance / Rejection Criteria

#### 4.8. UNITS

See analysis chapter for details related to units used for the different variables and calculations.

In case of collection of variables with non-SI units (e.g. pounds instead to kilograms), conversion of such data into SI units (and vice versa) will be ensured and both results will be reported for the full set of available subjects next to each other in the interim/annual and/or final reports.

### 4.9. CALCULATIONS AND TRANSFORMATIONS

Distances between times and differences between score results will be calculated. For full details of variables used for calculations and the creation of new variables based on these calculations, see analysis chapter.

### 4.10. ASSUMTIONS

In case of deviation from assumptions (e.g. normality), non-parametric methods will be used for analysis. No transformation of such data will be performed.

### 5. Population and Progress

#### 5.1. ANALYSIS POPULATION

It is expected, that during this clinical investigation only one population for Tibia will exist and all subjects will be analyzed "Per Protocol" (PP). However, it cannot be fully avoided that in theory subjects might need to be excluded from the PP population. In this occasion, there will be two groups being fully analyzed to ensure transparency and avoid bias.

The groups are defined as follows:

### • Intent-to Treat Population

The Intent-to-Treat (ITT) Population is defined to be all enrolled subjects. An enrolled subject is a subject that has signed informed consent, all screening procedures have been successfully completed, is eligible and can receive treatment. The ITT population will not be analyzed for the annual reports and will only be included in the final report.

### • Per Protocol Population

The Per Protocol (PP) Population is defined to be all subjects in the ITT Population with no major protocol violations. The protocol violations that will exclude a subject are as follows:

- The subject does not receive the T2 Alpha Tibia Nail
- The subject does not meet all eligibility criteria
- The subject has a protocol violation that is considered likely to affect subject outcomes.

After the clinical investigation has been completed, a review of the data will be conducted to determine which subjects are to be excluded from the PP population.

The following tables will be created for interim/annual and final reports related to the clinical investigation populations and progress:

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan |
|---|---|---|
| All Forms - Overview & Progres | s Report | |
| Counting of available subjects Subject Population by Site (Variable(s): SITENUM; SUBID) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of available subjects Subject Population by Visit (Variable(s): SITENUM; SUBID; VISITDT) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of available subjects Subject Population by Visit and by Site (Variable(s): SITENUM; SUBID; VISITDT) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |

Table 5.1: Populations and Progress Tables List

### 5.2. ELIGIBILITY

A subject is defined as eligible if all inclusion and exclusion criteria are fulfilled as it is described in the protocol. For details see CIP.

For tables to be created for the interim/annual and final reports, see chapter 6.2 and tables list 6.2.2.

### 5.3. WITHDRAWAL / FOLLOW-UP

If, during the clinical investigation, a subject must be prematurely withdrawn from clinical investigation, procedures are outlined in the CIP. These procedures should not interfere with the initiation of any new treatments that are necessary to treat a subject's condition. Information on all withdrawn subjects will be documented.

The following tables will be created for interim/annual and final reports related to the numbers of withdrawn subjects (if any):

| Evaluation | Level of | Analysis Plan |
|---|---|---|
| Variable / Question | Measurement | Anarysis I fan |
| All Forms - Overview & Progres | s Report | |
| Counting of withdrawn subjects Number of Subjects Withdrawn by Site (Variable(s): SITENUM; COMPPROT; PRIMRSN) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of withdrawn subjects Number of Subjects Withdrawn by Site by Visit (Variable(s): SITENUM; COMPPROT; PRIMRSN; VISITDT) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Comments related to Reasons for Subjects Withdrawn (Variable(s): RSNSPF) | Text, String | Listing of reasons for subjects being excluded by subject code/ID |

Table 5.3: Withdrawal Tables List

### 5.4. ADHERENCE AND CIP DEVIATIONS

Any CIP deviations will be listed in the interim/annual and final reports. It is optional to describe this chapter in free text or present it in a tabulated format.

### 6. Analysis

The following tabulated analysis plan reflects this approach and specifies the variables characteristics (quantitative or qualitative) in detail together with the related analysis strategy. This also includes calculation and summaries based on primary elements and the required analysis.

In addition, it will be defined in the text or directly in the tables below, if the variable must be included in an interim/annual report (IR) and/or in the final report (FR).

### 6.1. HARMS AND SAFETY

Categorization and definitions of (Serious-, Unanticipated-) Adverse Device Effects, (Serious-) Incidents are given in the CIP.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| Adverse Events / Incidents | | | IR | FR | N/A |
| Device-Related Adverse Event / Incident (Variable(s): AEEVENT; AEOTHER) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of other Events/Incidents. | X | X | |
| Describe the AE/Incident<br>(Variable(s): AEDESCRP) | Qualitative, nominal | Listing of other<br>Events/Incidents Description. | | | X |
| Unanticipated Adverse Device<br>Event?<br>(Variable(s): AEUADE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Severity<br>(Variable(s): AESEVER) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Describe Treatment:<br>(Variable(s): ACTTREAT) | Qualitative, nominal | Listing of Treatment Description. | | | X |
| Action Taken (Variable(s): ACTNONE; ACTMEDS; ACTSURG; ACTLABOT; ACTSHORT; ACTPROHS; ACTOTHER; ACTOTHSP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given Other specifications. | | | X |
| AE Resolution<br>(Variable(s): AERESOLV) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Outcome<br>(Variable(s): AEONWOTR;<br>AEONWTTR; AEREWOTR;<br>AEREWTTR; AETEDISB;<br>AEPERMD; AESUEXP) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Creation of variable Number of Adverse Device Effects by Site (Variable(s): AEEVENT; SITENUM) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Creation of variable Number of Adverse Device Effects per Subject and Site (Variable(s): AEEVENT; SITENUM; SUBID) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Creation of variable Number of<br>Adverse Device Effects by Visit<br>(Variable(s): AEEVENT; VISNAME) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |

Table 6.1: Adverse Events / Incidents Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| Reoperation | Reoperation | | | FR | N/A |
| Type of Procedure (Variable(s): TOPAMP; TOPDYNA; TOPIMPREM; TOPIRDEB; TOPRTAINTFIX; TOPINTSPF; TOPREVARTH; TOPARTHSPF; TOPRTAEXTFIX; TOPEXTSPF; TOPOTH; TOPOTHSPF) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listings of implant specifications. | X | X | |
| Reason(s) for Reoperation (Variable(s): DELUNION; IATRFRAC; IMPBRAK; IMPLFAIL; IMPLOOS; INFEC; MALILGN; MALUNI; NECRS; NONUNIO; PAIN; REOPOTH; REOPOTHSPF) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listings of other specifications. | X | X | |

Table 6.2: Reoperation Tables List

### 6.2. BASELINE CHARACTERISTICS

| Evaluation<br>Variable / Question | Level of Measurement | ment Analysis Plan | | Inclusion | |
|---|---|---|---|---|---|
| Pre-Operative Visit Form – Sub<br>Criteria | ject Eligibility – | Inclusion & Exclusion | IR | FR | N/A |
| Note: Inclusion and exclusion criteria wil fulfilled the inclusion criteria). | ll be checked during r | monitoring and reported by a state | ement (e | e.g. all s | ubjects |
| Inclusion Criteria Questions<br>(Variable(s): INCLA; INCLB; INCLC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Exclusion Criteria Questions<br>(Variable(s): EXCLA; EXCLB) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |

Table 6.2.1: Pre-Operative Visit Form - Subject Eligibility – Inclusion & Exclusion Criteria
Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| Pre-Operative Visit Form - Sub | | ics | IR | FR | N/A |
| Creation of variable Age [years] Difference between Date of Surgery [dd.mm.yyyy] and Date of Birth/DOB [dd.mm.yyyy] in [ years ] (Variable(s): BIRTHDT; VISITDT; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | х | |
| Gender<br>(Variable(s): GENDER) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Race<br>(Variable(s): AMERIND; ASIAN;<br>BLKAFR; NATHAW; CAUS;<br>RACEOTH; RACEOTHR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |
| Height [captured in inches or cm] In the analysis, all values will be reported in inches and cm next to each other. (Variable(s): HGHTM) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% | | | X |

| | | confidence interval for mean,<br>Shapiro-Wilk Test. | | | |
|---|---|---|---|---|---|
| Weight [captured in lbs or kg] In the analysis, all values will be reported in lbs and kg next to each other. (Variable(s): WEIGHTKG) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | Х |
| Body Mass Index [kg/m²]<br>(Variable(s): BMI) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |

Table 6.2.2: Pre-Operative Visit Form - Subject Demographics Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | |
|---|---|---|---|---|---|
| Pre-Operative Visit Form - Cui | rent Relevant M | <b>Iedical Conditions</b> | IR | FR | N/A |
| Current Relevant Medical<br>Conditions (Variable(s): CURCOND;<br>CONDSPC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |

Table 6.2.3: Pre-Operative Visit Form - Current Relevant Medical Conditions

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| <b>Pre-Operative Visit Form – Sub</b> | ject Evaluation | | IR | FR | N/A |
| Tobacco Use:<br>(Variable(s): TOBCCO) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Corticosteroids Taking:<br>(Variable(s): CORTICO) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Affected (Study) Tibia<br>(Variable(s): AFFCTIB) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Fracture Classification:<br>(Variable(s): FRUCLS) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Mechanism of Injury:<br>(Variable(s): MECHINJ; OTHSPC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |
| Primary Indication:<br>(Variable(s): PRIMIND) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |
| Previous History of Surgery to the<br>Affected Tibia<br>(Variable(s): PREVHIST) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | | X | |
| Procedure 1<br>(Variable(s): PROCNM1) | Text, String | | | | X |

| | T | T | 1 | | 1 |
|---|---|---|---|---|---|
| Procedure Date 1<br>(Variable(s): PROCDT1) | Quantitative,<br>ratio<br>Date/Time | Listing of comments and dates together identified by subject code/ID | | | X |
| Procedure 2 (Variable(s): PROCNM2) | Text, String | Listing of comments and | | | X |
| Procedure Date 2<br>(Variable(s): PROCDT2) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Procedure 3 (Variable(s): PROCNM3) | Text, String | Listing of comments and | | | X |
| Procedure Date 3<br>(Variable(s): PROCDT3) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Procedure 4 (Variable(s): PROCNM4) | Text, String | Listing of comments and | | | X |
| Procedure Date 4<br>(Variable(s): PROCDT4) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Previous History of Surgery to the<br>Contralateral Tibia<br>(Variable(s): PREVHISTCONTR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | | X | |
| Procedure 1 (Variable(s): CONTRPROCNM1) | Text, String | Listing of comments and | | | X |
| Procedure Date 1<br>(Variable(s): CONTRPROCDT1) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Procedure 2 (Variable(s): CONTRPROCNM2) | Text, String | Listing of comments and | | | X |
| Procedure Date 2<br>(Variable(s): CONTRPROCDT2) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Procedure 3 (Variable(s): CONTRPROCNM3) | Text, String | Listing of comments and | | | X |
| Procedure Date 3 (Variable(s): CONTRPROCDT3) | Quantitative,<br>ratio<br>Date/Time | dates together identified by subject code/ID | | | X |
| Procedure 4 (Variable(s): CONTRPROCNM4) | Text, String | Listing of comments and | | | X |
| Procedure Date 4 (Variable(s): CONTRPROCDT4) | Quantitative, ratio Date/Time | dates together identified by subject code/ID | | | X |
| Creation of variable Number of previous history of surgery to the Affected Tibia by Subject (Variable(s): PROCNM1; PROCNM2; PROCNM3; PROCNM4) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Creation of variable Number of previous history of surgery to the Contralateral Tibia by Subject (Variable(s): CONTRPROCNM1; CONTRPROCNM2; CONTRPROCNM3; CONTRPROCNM4) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Weight Bearing (Variable(s): WEIGTBEAR) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Weight Bearing Specification<br>(Variable(s): WEIGTSPC) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| External Support Prior to the Tibia<br>Fracture<br>(Variable(s): EXTRSUPP) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |

Table 6.2.4: Pre-Operative Visit Form – Subject Evaluation Tables List

| Evaluation | Level of | Analysis Plan | | | |
|---|---|---|---|---|---|
| Variable / Question | Measurement | • | - | nclusio | |
| Pre-Operative Visit Form – SF- | 36 Score (post fi | acture, prior to | IR | FR | N/A |
| surgery) | | | 110 | 110 | 1 1/11 |
| In general, would you say your | Qualitative, | Proportions, frequencies, | | | |
| health is | nominal | column and row totals, | | | X |
| (Variable(s): GH01_RESPONSE) Compared to one year ago, how | | missing proportion (if any). | - | | |
| would you rate your health in | Qualitative, | Proportions, frequencies, | | | |
| general now? | nominal | column and row totals, | | | X |
| (Variable(s): HT RESPONSE) | | missing proportion (if any). | | | |
| Vigorous activities, such as running, | | Proportions, frequencies, | | | |
| lifting heavy objects, participating in | Qualitative, | column and row totals, | | | X |
| strenuous sports | nominal | missing proportion (if any). | | | 1 |
| (Variable(s): PF01 RESPONSE) Moderate activities, such as moving a | | 31 1 ( 3) | | | |
| table, pushing a vacuum cleaner, | Qualitative, | Proportions, frequencies, | | | |
| bowling, or playing golf | nominal | column and row totals, | | | X |
| (Variable(s): PF02 RESPONSE) | nommar | missing proportion (if any). | | | |
| | Qualitation | Proportions, frequencies, | | | |
| Lifting or carrying groceries (Variable(s): PF03 RESPONSE) | Qualitative, | column and row totals, | 1 | | X |
| ( variable(s), 1 ros_Response) | nommai | missing proportion (if any). | | | |
| Climbing several flights of stairs | Qualitative, | Proportions, frequencies, | 1 | | |
| (Variable(s): PF04_RESPONSE) | nominal | column and row totals, | 1 | | X |
| | | missing proportion (if any). | | | |
| Climbing one flight of stairs | Qualitative, | Proportions, frequencies, column and row totals, | | | X |
| (Variable(s): PF05_RESPONSE) | nominal | missing proportion (if any). | | | Α |
| | | Proportions, frequencies, | | | |
| Bending, kneeling, or stooping | Qualitative, | column and row totals, | | | X |
| (Variable(s): PF06_RESPONSE) | nominal | missing proportion (if any). | | | |
| Walking more than a mile | Qualitative, | Proportions, frequencies, | | | |
| (Variable(s): PF07 RESPONSE) | nominal | column and row totals, | | | X |
| (variable(s):11 ov_1ezst sit(sz) | Понина | missing proportion (if any). | | | |
| Walking several hundred yards | Qualitative, | Proportions, frequencies, | | | X |
| (Variable(s): PF08_RESPONSE) | nominal | column and row totals, missing proportion (if any). | | | A |
| | | Proportions, frequencies, | | | |
| Walking one hundred yards | Qualitative, | column and row totals, | | | X |
| (Variable(s): PF09_RESPONSE) | nominal | missing proportion (if any). | | | |
| Bathing or dressing yourself | Qualitative, | Proportions, frequencies, | | | |
| (Variable(s): PF10 RESPONSE) | nominal | column and row totals, | | | X |
| ` '/ = / | Понина | missing proportion (if any). | | | |
| Cut down the amount of time you | Qualitative, | Proportions, frequencies, | | | 37 |
| spent on work or other activities (Variable(s): RP01 RESPONSE) | nominal | column and row totals, missing proportion (if any). | | | X |
| Accomplished less than you would | | Proportions, frequencies, | | | |
| like | Qualitative, | column and row totals, | | | X |
| (Variable(s): RP02 RESPONSE) | nominal | missing proportion (if any). | <u>L</u> | | L - |
| Were limited in the kind of work or | Qualitative, | Proportions, frequencies, | | | |
| other activities | nominal | column and row totals, | | | X |
| (Variable(s): RP03_RESPONSE) | | missing proportion (if any). | 1 | | |
| Had difficulty performing the work | | Proportions fraguesias | 1 | | |
| or<br>other activities (for example, it took | Qualitative, | Proportions, frequencies, column and row totals, | 1 | | X |
| extra effort) | nominal | missing proportion (if any). | 1 | | '` |
| (Variable(s): RP04_RESPONSE) | | Grapation (it will). | | | |
| Cut down the amount of time you | Qualitativa | Proportions, frequencies, | | | |
| spent on work or other activities | Qualitative, nominal | column and row totals, | 1 | | X |
| (Variable(s): RE01_RESPONSE) | nommai | missing proportion (if any). | | | |
| Accomplished less than you would | Qualitative, | Proportions, frequencies, | 1 | | |
| like | nominal | column and row totals, | 1 | | X |
| (Variable(s): RE02 RESPONSE) Did work or other activities less | | missing proportion (if any). Proportions, frequencies, | | | |
| carefully than usual | Qualitative, | column and row totals, | 1 | | X |
| (Variable(s): RE03 RESPONSE) | nominal | missing proportion (if any). | 1 | | 1 |

| During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01_RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP01_RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): WH04_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, | x x x x x x |
|---|---|
| emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, Pominal During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you feel downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X X X X |
| your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you feel tdownhearted and depressed? (Variable(s): MH04 RESPONSE) Did you feel worn out? Qualitative, nominal Column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). | X X X X |
| family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) | X X X X |
| Groups? (Variable(s): SF01 RESPONSE) | x x x x |
| Oualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | x x x x |
| How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X X X X |
| Column and row totals, wissing proportion (if any). | X X X X |
| During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) | X<br>X<br>X |
| did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion, frequencies, column and row totals, missing pro | X<br>X<br>X |
| work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? Qualitative, nominal Column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). | X<br>X<br>X |
| the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Qualitative, nominal Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X<br>X<br>X |
| Oualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Did you feel full of life? (Variable(s): VT01_RESPONSE) | X |
| Column and row totals, missing proportion (if any). | X |
| Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you felt worn out? Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Column and row totals, missing proportion (if any). | X |
| (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | |
| that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | |
| that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | |
| Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Column and row totals, missing proportion (if any). | X |
| Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | 1 21 |
| Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion, frequencies, column and row totals, missing proportion, frequencies, column and row totals. | |
| Column and row totals, missing proportion (if any). | |
| Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? Missing proportion (if any). | X |
| depressed?<br>(Variable(s): MH04 RESPONSE) Qualitative,<br>nominal column and row totals,<br>missing proportion (if any). Did you feel worn out? Qualitative,<br>Qualitative, Proportions, frequencies,<br>column and row totals | |
| Column and row totals, missing proportion (if any). | |
| (Variable(s): MH04_RESPONSE) missing proportion (if any). Did you feel worn out? Qualitative, Qualitative, column and row totals | X |
| Did you leef worli out: Qualitative, column and row totals | + |
| | X |
| (Variable(s): VT03_RESPONSE) nominal continuation totals, missing proportion (if any). | Λ |
| Proportions frequencies | |
| Have you been nappy? Quantative, | X |
| (Variable(s): MH05_RESPONSE) nominal continuation row totals, missing proportion (if any). | |
| Did you feel tired? Qualitative, Proportions, frequencies, | |
| (Variable(s): VT04 RESPONSE) nominal Column and row totals, | X |
| missing proportion (if any). | $\bot$ |
| During the past 4 weeks, how much | |
| of the time has your physical health | |
| or emotional problems interfered with Qualitative, column and row totals, | X |
| your social activities (like visiting nominal nominal missing proportion (if any). | Α |
| friends, relatives, etc.)? | |
| (Variable(s): SF02_RESPONSE) | |
| I seem to get sick a little easier than Ouglitative Proportions, frequencies, | |
| other people column and row totals, | X |
| (Variable(s): GH02 RESPONSE) missing proportion (if any). | |
| I am as healthy as anybody I know Qualitative, Proportions, frequencies, | 37 |
| (Variable(s): GH03_RESPONSE) Qualitative, nominal column and row totals, missing proportion (if any). | X |
| Proportions frequencies | + |
| 1 expect my nealth to get worse Qualitative, column and row totals | X |
| (Variable(s): GH04_RESPONSE) nominal contains and row totals, missing proportion (if any). | '` |
| Proportions fraguancies | |
| (Variable(s): GH05 RESPONSE) quantative, column and row totals, | X |
| missing proportion (if any). | |
| Case summary with number | |
| and percentage of valid | |
| Characteristics cases/values, missing | |
| Physical Functioning<br>(Variable(s): PFSCORE) Quantitative,<br>ratio cases/values (if any) and total<br>cases/values. X | |
| (variable(s): PFSCORE) ratio cases/values. Mean, median, interquartile | 1 |
| range, maximum, minimum, | |
| standard deviation, 95% | |

| | | 0.1 | 1 | | 1 |
|---|---|---|---|---|---|
| | | confidence interval for mean,<br>Shapiro-Wilk Test. | | | |
| Role Physical<br>(Variable(s): RPSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, | X | X | |
| Bodily Pain (Variable(s): BPSCORE) | Quantitative, ratio | Shapiro-Wilk Test. Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| General Health<br>(Variable(s): GHSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | Х | |
| Vitality<br>(Variable(s): VTSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Social Functioning<br>(Variable(s): SFSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | X | |
| Role Emotional<br>(Variable(s): RESCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Mental Health<br>(Variable(s): MHSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, | Х | Х | |

| | | standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | |
|---|---|---|---|---|
| Total Physical Score<br>(Variable(s): PCSSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | X |
| Total Mental Score<br>(Variable(s): MCSSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X |

Table 6.2.5: Pre-Operative Visit Form – SF-36 Score (post fracture, prior to surgery) Tables List

### 6.3. INTRA-OPERATIVE CHARACTERISTICS

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| <b>Operative Visit – Operative Pro</b> | cedure | | IR | FR | N/A |
| Date of Surgery: (Variable(s): VISITDT; VISNAME) | Date/Time | Listing the first and last<br>surgery in the report text to<br>describe from which date to<br>which date subjects were<br>operated. | | X | |
| Date of Admission: (Variable(s): ADMINDT; VISNAME) | Date/Time | None | | | X |
| Date of Discharge: (Variable(s): DISCHRDT; VISNAME) | Date/Time | None | | | X |
| Creation of variable Difference between Date of Admission [dd.mm.yyyy] and Date of Surgery [dd.mm.yyyy] in days (Variable(s): ADMINDT; VISITDT; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Surgery Start Time (24 hour clock): (Variable(s): SURGSTTM) | Date/Time | None | | | X |
| Surgery Stop Time (24 hour clock): (Variable(s): SURGSPTM) | Date/Time | None | | | X |
| Difference between Surgery Start Time and Surgery Stop Time in hh:mm (Variable(s): SURGSTTM; SURGSPTM) | Quantitative,<br>ratio<br>Date/Time | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | х | |
| Amount of Blood Infused<br>(Variable(s): BLOODINF) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing | | X | |

| | | cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | |
|---|---|---|---|---|
| Type of Anesthesia: (Variable(s): TYPANEST) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Were there any technical difficulties<br>during surgery?<br>(Variable(s): SURGDIFF;<br>SURGDESC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | X | X |
| Were any concomitant procedure<br>done during surgery?<br>(Variable(s): CONPROC;<br>CONPROCD) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | X | X |

Table 6.3.1: Operative Visit – Surgical Procedure Tables List

| Evaluation | Level of | A l DI | т. | 1 | |
|---|---|---|---|---|---|
| Variable / Question | Measurement | Analysis Plan | Inclusion | | on |
| <b>Operative Visit – Implant Speci</b> | fication and Loc | king Information | IR | FR | N/A |
| Nail Reference Number (xxxx/xxxx): (Variable(s): REFNUM) | Qualitative,<br>nominal | None, used to populate nail details into database | | | X |
| Approach<br>(Variable(s): APPRCH) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Proximal Locking Mode<br>(Variable(s): PROXLOCMD) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| If Static Proximal Locking Mode<br>(Variable(s): PRXOBLSTLSCR;<br>PRXOBLANGSC; DISOBLSTLSCR;<br>DISOBLANGLSCR; OBLSTLSCR;<br>MLSTLSCR; MLSTANGLSCR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Distal Locking Screws (Variable(s): PROMLSTLSCR; PROMLANGLSCR; DISMLSTNLSCR; DISMLANGLSCR; APSTNLSCR; APANGLSCR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Was the Distal Targeting Device used? (Variable(s): DISTTARGT) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Was an End Cap used?<br>(Variable(s): ENDCAP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| If yes, check which length of End<br>Cap was used<br>(Variable(s): ENDCAPLENTH) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |

Table 6.3.2: Operative Visit – Implant Specification and Locking Information

### 6.4. EARLY POST-OPERATIVE CHARACTERISTICS

N/A

### 6.5. POST-OPERATIVE CHARACTERISTICS

The analysis of the Postoperative data must be performed separately for each follow-up visit listed in table 4.4 in accordance to the following tables in this chapter. New Variables must be created individually for each follow-up visit.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| | Post-Operative Visit Form – Physical Exam | | | | |
| Date of Visit: | Date/Time | None | | | X |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of Visit [dd.mm.yyyy] In [ days ] (Variable(s): VISITID; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Is the subject weight bearing? (Variable(s): WEIGHTBEAR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Specify, Full or Partial (Variable(s): FULPART) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Is the subject using an external support? (Variable(s): EXTRSUPP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Has the bone consolidated (consider weight-bearing, pain and imaging)? (Variable(s): BONECONS; EXPLN) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given explanations. | X | X | |

Table 6.5.1: Post-Operative Visit Form – Physical Exam Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| Post-Operative Visit Form – SF | | | IR | FR | N/A |
| In general, would you say your<br>health is<br>(Variable(s): GH01 RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | Х |
| Compared to one year ago, how<br>would you rate your health in<br>general now?<br>(Variable(s): HT RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Vigorous activities, such as running,<br>lifting heavy objects, participating in<br>strenuous sports<br>(Variable(s): PF01 RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf (Variable(s): PF02 RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Lifting or carrying groceries<br>(Variable(s): PF03_RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Climbing several flights of stairs (Variable(s): PF04_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Climbing one flight of stairs<br>(Variable(s): PF05_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Bending, kneeling, or stooping<br>(Variable(s): PF06_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Walking more than a mile<br>(Variable(s): PF07_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Walking several hundred yards<br>(Variable(s): PF08_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |

| Nalking one hundred yards (Variable(s): PF09 RESPONSE) nominal column and row totals, missing proportion (if any). Bathing or dressing yourself (Variable(s): PF10 RESPONSE) nominal row totals, missing proportion (if any). Cut down the amount of time you spent on work or other activities (Variable(s): RP01 RESPONSE) (Variable(s): RP02 RESPONSE) (Variable(s): RP02 RESPONSE) (Variable(s): RP02 RESPONSE) (Variable(s): RP02 RESPONSE) (Variable(s): RP03 RESPONSE) (Variable(s): RP03 RESPONSE) (Variable(s): RP03 RESPONSE) (Variable(s): RP04 RESPONSE) (Variable(s): RP | | T | | |
|---|---|---|---|---|
| Rathing or dressing yourself (Variable(s): PF09 RESPONSE) Oualitative, comminal missing proportion (if any). Oualitative, comminal command or words or dear activities (Variable(s): PR01 RESPONSE) Oualitative, comminal command or words or dear activities (Variable(s): RP03 RESPONSE) Martin or other activities (Variable(s): RP03 RESPONSE) Had difficulty performing the work or other activities (Variable(s): RP03 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP03 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP03 RESPONSE) Diffigure the past 4 weeks, to what cutent has your portunal social activities with family, friends, neighbors, or groups? (Variable(s): RP03 RESPONSE) During the past 4 weeks, to what cutent has your normal soutied pain interfered with your normal work (including both work outside the home and housework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has your normal soutied pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has youn both sousework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has youn housework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has youn housework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has youn housework)? (Variable(s): RP00 RESPONSE) During the past 4 weeks, to what cutent has youn formal more volument and row totals, missing proportion (if any). **Column and row totals, missin | Walking one hundred vards | Qualitative. | Proportions, frequencies, | |
| Bathing or dressing yourself (Variable(s): PF10 RISPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP01 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP02 RESPONSE) Cut down the amount of time you would like (Variable(s): RP02 RESPONSE) Cut down the amount of time you would like (Variable(s): RP03 RESPONSE) Cut down the amount of time you would like (Variable(s): RP03 RESPONSE) Cut down the amount of time you would like (Variable(s): RP04 RESPONSE) Cut down the amount of time you would like (Variable(s): RP04 RESPONSE) Cut down the amount of time you would like (Variable(s): RP04 RESPONSE) Did work or other activities (Portification with a comminal may be a lot of energy of Variable(s): RP04 RESPONSE) Town much bodily pain have you had during the past 4 weeks, to mominal much finely your normal work (including both work cutside the home and housework)? (Variable(s): RP01 RESPONSE) Town much bodily pain have you had during the past 4 weeks, to mominal much finely your normal work (including both work cutside the home and housework)? (Variable(s): RP02 RESPONSE) Town much bodily pain have you had during the past 4 weeks, to mominal much finely pain have you had work (including both work cutside the home and housework)? (Variable(s): RP01 RESPONSE) Tave you felt full of life? (Variable(s): VT01 RESPONSE) Tave you felt full of life? (Variable(s): MF01 RESPONSE) Tave you felt and mad peaceful? (Variable(s): MF01 RESPONSE) Did you have a lot of energy? (Variable(s): MF02 RESPONSE) Did you have a lot of energy? (Variable(s): MF03 RESPONSE) Did you felt would continue the dumps that nothing could cheer you up (Variable(s): MF01 RESPONSE) Did you felt and mad peaceful? (Variable(s): MF01 RESPONSE) Did you felt would continue the full of life? (Variable(s): MF01 RESPONSE) Did you felt would continue the full of life? (Variable(s): MF01 RESPONSE) Did you felt would continue the full of life? (Variable(s): MF01 RESPONSE | | 1 2 | | X |
| odulmatory of versus groups of groups groups of versus groups of groups of versus groups of | (+ 4214616(8): 11 05 _14281 01 (82) | 1101111111 | | |
| (Variable(s): P10 RESPONSE) Outloam the amount of time you spent on work or other activities (Variable(s): RP02 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP04 RESPONSE) Oualitative, nominal Were limited in the kind of work or other activities (Variable(s): RP04 RESPONSE) Oualitative, nominal Were limited in the kind of work or other activities (Variable(s): RP04 RESPONSE) Oualitative, nominal Wariable(s): RP03 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RP04 RESPONSE) Did work or other activities with family, friends, neighbors, or groups? (Variable(s): RP03 RESPONSE) How much bodily pain have you had during the past 4 weeks, to whate extent has your physical health or mominal mover (including both work outside the hone and housework)? (Variable(s): RP01 RESPONSE) Did you feel full of life? (Variable(s): RP01 RESPONSE) Did you feel full of life? (Variable(s): RP03 RESPONSE) Did you feel full of life? (Variable(s): RP03 RESPONSE) Did you feel full of life? (Variable(s): RP04 RESPONSE) Did you feel full of life? (Variable(s): RP05 RESPONSE) Did you feel full of life? (Variable(s): RP07 RESPONSE) Did you feel full of life? (Variable(s): RP08 RESPONSE) Did you feel full of life? (Variable(s): RP09 RESPONSE) Did you feel full of life? (Variable(s): RP09 RESPONSE) Did you feel work or outside the hone and houseward and you feel so down in the dumps that nothing could chear you up. (Variable(s): RP09 RESPONSE) Did you feel work or outside the hone and houseward and you feel so down in the dumps that nothing | Bathing or dressing yourself | Oualitative. | | |
| Cut down the amount of time you spent on work or other activities (Variable(s)-RP01 RESPONSE) Accomplished less than you would like (Variable(s)-RP02 RESPONSE) Had difficulty performing the work or other activities (Variable(s)-RP03 RESPONSE) Had difficulty performing the work or other activities (for example, it took cut and the you spent on work or other activities (Variable(s)-RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s)-RP04 RESPONSE) Accomplished less than you would like (Variable(s)-RP03 RESPONSE) Did work or other activities (Variable(s)-RP03 RESPONSE) How much bodity pain have you had during the past 4 weeks, to what extent has your physical health or comotional problems interfered with your normal work (including both work outside the home and housework)? (Variable(s)-RP03 RESPONSE) Did you feel full of life? (Variable(s)-RP03 RESPONSE) Did you feel full of life? (Variable(s)-RP03 RESPONSE) Did you feel full of life? (Variable(s)-RP03 RESPONSE) Did you feel full of life? (Variable(s)-RP03 RESPONSE) Did you feel full of life? (Variable(s)-RP03 RESPONSE) Did you have a lot of energy? (Variable(s)-RP03 RESPONSE) Did you feel fall of life? (Variable(s)-RP03 RESPONSE) Did you feel fall of life? (Variable(s)-RP03 RESPONSE) Did you feel foul of life? (Variable(s)-RP03 RESP | | | | X |
| spent on work or other activities (Variable(s): RPO1 RESPONSE) Accomplished less than you would like (Variable(s): RPO2 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RPO3 RESPONSE) Had difficulty performing the work or other activities (for example, it took extra effort) (Variable(s): RPO4 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RPO4 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RPO4 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): REO1 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): REO2 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): REO2 RESPONSE) Did work or other activities less carefully than usual (Variable(s): REO2 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SPO1 RESPONSE) During the past 4 weeks? (Variable(s): PRO2 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): VTO1 RESPONSE) Did you feel full of life? (Variable(s): WTO1 RESPONSE) Have you feel so down in the dumps attained and one wood to tals, moising proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequenc | <u> </u> | | | |
| spent on work or other activities (Variable(s): PRO12_RESPONSE) Accomplished less than you would like (Variable(s): RP02_RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03_RESPONSE) Had difficulty performing the work or other activities (for example, it took extra effort) (Variable(s): RP04_RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04_RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04_RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP02_RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04_RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04_RESPONSE) Did work or other activities less carefully than usual (Variable(s): RP03_RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): RP01_RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SP01_RESPONSE) During the past 4 weeks, tow much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP01_RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): MP01_RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): MP01_RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): MP01_RESPONSE) During the past 4 weeks, to mominal missing proportion (if any). Proportions, frequenc | | Qualitative, | | 37 |
| Accomplished less than you would like (Variable(s): RP02 RESPONSE) Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) (Variable(s): RP03 RESPONSE) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP02 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RP03 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RP03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): RP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework?) (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WT01 RESPONSE) Did you feel work out of energy? (Variable(s): MH01 RESPONSE) Did you feel work out of energy? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): WH04 RESPONSE) Did you feel worn out? (V | | 1 2 | | X |
| like (Variable(s): RP02 RESPONSE) Were finited in the kind of work or other activities (Variable(s): RP03 RESPONSE) Had difficulty performing the work or other activities (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities (Variable(s): RE02 RESPONSE) Did work or other activities (Variable(s): RE03 RESPONSE) Did work or other activities (Variable(s): RE03 RESPONSE) Did work or other activities (Variable(s): RE03 RESPONSE) Did work or other activities (Variable(s): RE03 RESPONSE) How much bodity pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): PP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you feel to down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you feet fact am and peaceful? (Variable(s): HM03 RESPONSE) Did you feet fact than and excentil? (Variable(s): WH03 RESPONSE) Have you feet call and peaceful? (Variable(s): WH03 RESPONSE) Did you feet fact than and generated and depressed? (Variable(s): HM04 RESPONSE) Did you feet foll of life? (Variable(s): WH03 RESPONSE) Did you feet fact dum and generated and depressed? (Variable(s): HM04 RESPONSE) Did you feet foll of life? (Variable(s): WH03 RESPONSE) Did you feet foll of life? (Variable(s): WH03 RESPONSE) Did you have a lot of energy? (Variable(s): HM04 RESPONSE) Did you feet foll of life? (Variable(s): WH03 RESPONSE) Did you feet foll of life? (Variable(s): WH04 RESPONSE) Did you feet foll of energy? (Variable(s): WH04 | | | | |
| Were fimited in the kind of work or other activities (CVariable(s): RP02 RESPONSE) More factivities (for example, it took other activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Qualitative, nominal Qualitative, | | Qualitative, | | 37 |
| Were limited in the kind of work or other activities (Variable(s): RP03 RESPONSE) National Management of the activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RP04 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RP04 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RP04 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RE02 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RE02 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): RE03 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): SF01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): BP01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): BP01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WT01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WT01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WT01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WT01 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WH02 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WH03 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WH03 RESPONSE) Qualitative, nominal missing proportion (if any). Yamabele(s): WH04 RESPONSE) Qualitative, nominal missing proportion (if any). | | | | X |
| other activities (Variable(s), RP03 RESPONSE) Had difficulty performing the work or other activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or comotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): RF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, to much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP01 RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Did you feel to down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Did you have a lot of energy? (Variable(s): WH02_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you nevel downhearted and depressed? (Variable(s): WH03_RESPONSE) Did you nevel downhearted and depressed? (Variable(s): WH03_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH03_RESPONSE) Qualitative, nominal Did you feel to man peaceful? (Variable(s): WH04_RESPONSE) Qualitative, nominal Did you have a lot of energy? (Variable(s): WH04_RESPONSE) Qualitative, nominal Did you feel to man peaceful? (Variable(s): WH04_RESPONSE) Qualitative, nominal Did you feel worn out? (Variable(s): WH04_R | | | | |
| omeinal materior volusis. A continual and row totals. The column and row to | | Qualitative, | | 37 |
| Had difficulty performing the work or ofter activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or nother activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, now much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WH01 RESPONSE) Have you been very nervous? (Variable(s): WH01 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): WH01 RESPONSE) Have you felt calm and peaceful? (Variable(s): WH02 RESPONSE) Did you have a lot of energy? (Variable(s): WH03 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you feel fel with or centre of the peace of | | | | |
| or other activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or comotional problems interfered with your normal social activities with family, friends, neighbors, or mominal Work including both work outside the home and housework? (Variable(s): BP02 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): MF01 RESPONSE) Did you feel full of life? (Variable(s): MH01 RESPONSE) Have you been very nervous? (Variable(s): MH01 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH01 RESPONSE) Have you felt downhearted and depressed? (Variable(s): VT02 RESPONSE) Did you have a lot of energy? (Variable(s): WH01 RESPONSE) Did you have a lot of energy? (Variable(s): WH01 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you have a lot of energy? (Variable(s): WH04 RESPONSE) Did you feel worn out? (Variable(s): WH05 RESPONSE) Did you feel worn out? (Variable(s): WH05 RESPONSE) Did you feel worn out? (Variable(s): WH05 RESPONSE) Did you been happy? (Variable(s): WH05 RESPONSE) Did you been happy? (Variable(s): WH05 RESPONSE) | | | missing proportion (if any). | |
| other activities (for example, it took extra effort) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with your normal social activities with gour health or emotional problems interfered with your much bodily pain have you had did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WH01_RESPONSE) Have you been very nervous? (Variable(s): MH02_RESPONSE) Qualitative, nominal Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you feel full of life? (Variable(s): WH03_RESPONSE) Qualitative, nominal Accomplished less than you would in the dumps that nothing could cheer you up? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) | | | | |
| cutra effort) (Variable(s): RP04 RESPONSE) Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or camotional problems interfered wity your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, wo much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WH01_RESPONSE) Have you been very nervous? (Variable(s): MH02_RESPONSE) Did you have a lot of energy? (Variable(s): WH02_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel won out? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH05_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you | | Qualitative, | | v |
| Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Oualitative, nominal Oualitative, n | | | | |
| Cut down the amount of time you spent on work or other activities (Variable(s): RE01 RESPONSE) Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): MH01 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02 RESPONSE) Did you feel downhearted and depressed? (Variable(s): WT02 RESPONSE) Did you feel full own the dumps that nothing could cheer you up? (Variable(s): WT02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02 RESPONSE) Did you feel for control of the down and the down and row totals, missing proportion (if any). The column and row totals, missing proportion (if any). Wariable(s): WT02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02 RESPONSE) Did you feel worn out? (Variable(s): WT03 RESPONSE) Did you feel worn out? (Va | | | missing proportion (if any). | |
| spent on work or other activities (Variable(s): RE01_RESPONSE) Accomplished less than you would like (Variable(s): RE02_RESPONSE) Did work or other activities less carefully than usual vertent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SP01_RESPONSE) How much bodily pain have you had during the past 4 weeks, tow much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02_RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Did you feel dam and peaceful? (Variable(s): MH02_RESPONSE) Did you feel dam and peaceful? (Variable(s): MH03_RESPONSE) Did you feel dam and peaceful? (Variable(s): MH03_RESPONSE) Did you feel dam and peaceful? (Variable(s): MH03_RESPONSE) Did you feel dam and peaceful? (Variable(s): WH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WH04_RESPONSE) Did you feel worn out? (Variable(s): WH04_RESPONSE) Did you feel wouth out feel word out feel you feel | | 1 | Duran anti- una fina | + + - |
| column and row totals, missing proportion (if any). Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SP01 RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Have you been very nervous? (Variable(s): MH02 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you feel toll may be to down and power of the | | Qualitative, | | 37 |
| Accomplished less than you would like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside he home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WT01 RESPONSE) Have you been very nervous? (Variable(s): WH01 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you feel downhearted and depressed? (Variable(s): WT03_RESPONSE) Did you feel worn out? (Variable(s): WT04_RESPONSE) Did you feel worn out? | | 1 2 | | |
| like (Variable(s): RE02 RESPONSE) Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): RE07 RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP01 RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Have you been very nervous? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you feel down in the dumps that nothing could cheer you up? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): MH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you feel town out? (Variable(s): MH04 RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and r | | 1 | | + + - |
| nominal markey totals, yellow rotals and row totals, missing proportion (if any). Did work or other activities less carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you felt sod own in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you feel downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): WH04 RESPONSE) Did you feel worn out? (Variable(s): WH05 RESPONSE) Did you feel worn out? (Variable(s): WH05 RESPONSE) Did you feel worn out? (variable(s): WH05 RESPONSE) Did you feel worn ou | | Qualitative, | | 37 |
| Did work or other activities less carefully than usual (Variable(s): REO3 RESPONSE) | | 1 2 | | |
| carefully than usual (Variable(s): RE03 RESPONSE) During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, now much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): WT01_RESPONSE) Have you been very nervous? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): WT03_RESPONSE) Outlitative, nominal more votals, missing proportion (if any). The proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yamishle(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): WT03_RESPONSE) Did you feel worn out? (Variable(s): WT03_RESPONSE) Did you feel worn out? (Variable(s): WT03_RESPONSE) Availative, nominal Did you feel worn out? (Variable(s): WT03_RESPONSE) Did you feel worn out? (Variable(s): WH05_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and | | | | + + + - |
| Ouring the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? | | Qualitative, | | V |
| During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): WH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Pro | | nominal | | |
| extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Have you felt calm and peaceful? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Ave you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn our? (Variable(s): MH04_RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Yaminal proportion (if any). Yaminal proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any) | | | missing proportion (if any). | |
| emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01_RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01_RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02_RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): WT03_RESPONSE) Did you felt worn out? (Variable(s): WH05_RESPONSE) Did you felt worn out? (Variable(s): WH04_RESPONSE) Did you felt worn out? (Variable(s): WH05_RESPONSE) Qualitative, nominal Did you felt worn out? (Variable(s): WH05_RESPONSE) Qualitative, nominal Did you felt worn out? (Variable(s): WH05_RESPONSE) Qualitative, nominal Did you felt worn out? (Variable(s): WH05_RESPONSE) Qualitative, nominal Qualitative, nominal Droportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proporti | | | | |
| your normal social activities with family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01 RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you have a lot of energy? (Variable(s): WH03_RESPONSE) Did you have a lot of energy? (Variable(s): MH04 RESPONSE) Did you have a lot of energy? (Variable(s): MH04 RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you felt worn out? (Variable(s): MH04 RESPONSE) Did you felt worn out? (Variable(s): MH05_RESPONSE) Did you felt worn out? (Variable(s): MH04 RESPONSE) Did you felt worn out? (Variable(s): MH04 RESPONSE) Did you felt worn out? (Variable(s): MH05_RESPONSE) Did you felt worn out? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): MH05_RESPONSE) Did you felt worn out? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): MH05_RESPONSE) Did y | | | Decreations for manica | |
| family, friends, neighbors, or groups? (Variable(s): SF01 RESPONSE) How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Available(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): VT02_RESPONSE) Available(s): MH04_RESPONSE) Did you felt downhearted and depressed? (Variable(s): VT03_RESPONSE) Available(s): MH04_RESPONSE) Did you felt downhearted and depressed? (Variable(s): VT03_RESPONSE) Available(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): VT03_RESPONSE) Did you felt worn out? (Variable(s): VT03_RESPONSE) Available(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): VT03_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Proport | | Qualitative, | | V |
| Groups Charlabe(s): SF01 RESPONSE | | nominal | | A |
| Toportions (requencies, column and row totals, missing proportion (if any). Toportions (requencies, column and row totals, missing proportion (if any). | | | missing proportion (ii any). | |
| How much bodily pain have you had during the past 4 weeks? (Variable(s): BP01 RESPONSE) During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Did you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): WT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you fele worn out? (Variable(s): MH04_RESPONSE) Did you fele worn out? (Variable(s): WT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missin | | | | |
| Column and row totals, nominal Column and row totals, missing proportion (if any). | | | Proportions fraquencies | |
| Oualitative, nominal missing proportion (if any). Oualitative, nominal missing proportion (if any). | | Qualitative, | | |
| During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): MH04 RESPONSE) Did you feel town hout? (Variable(s): WH04 RESPONSE) Did you feel worn out? (Variable(s): WH05_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Did you feel worn out? (Variable(s): WH05_RESPONSE) Did you feel worn out? (Variable(s): WH05_RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | | nominal | | |
| did pain interfere with your normal work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH03_RESPONSE) Have you felt calm and peaceful? (Variable(s): WH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have felt downhearted and depressed? (Variable(s): WH04 RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). | | | imissing proportion (if any). | |
| work (including both work outside the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you have a lot of energy? (Variable(s): MH04_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Poportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row to | | | Proportions frequencies | |
| the home and housework)? (Variable(s): BP02 RESPONSE) Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, colu | | 1 2 | | X |
| Did you feel full of life? (Variable(s): VT01_RESPONSE) | | nominal | | |
| Did you feel full of life? (Variable(s): VT01_RESPONSE) Have you been very nervous? (Variable(s): MH01_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | | | initiality proportion (in unity). | |
| Column and row totals, missing proportion (if any). | | | Proportions, frequencies. | |
| Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | | | | X |
| Have you been very nervous? (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). | (variable(s): V101_RESPONSE) | nominal | | |
| (Variable(s): MH01_RESPONSE) Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02_RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Did you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you felt worn out? (Variable(s): WT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | п 1 | 0 11: -1 | | |
| Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | | | | |
| Have you felt so down in the dumps that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | (variable(s): MHUI_KESPONSE) | nominal | | |
| that nothing could cheer you up? (Variable(s): MH02 RESPONSE) Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Proportions, frequencies, column and row totals, missing proportion (if any). | Have you felt so down in the dumps | O1'4-4' | | |
| Wariable(s): MH02_RESPONSE nominal missing proportion (if any). | | ` ′ | | X |
| Have you felt calm and peaceful? (Variable(s): MH03_RESPONSE) Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | | nominal | | |
| Column and row totals, missing proportion (if any). Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). X | | Ovalit-ti- | | |
| Did you have a lot of energy? (Variable(s): VT02_RESPONSE) | | | | X |
| Did you have a lot of energy? (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | (Variable(s): MH03_RESPONSE) | nominal | | |
| (Variable(s): VT02_RESPONSE) Have you felt downhearted and depressed? (Variable(s): MH04_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). | Did you have a lat of any or 0 | Ovalit-ti- | | |
| Have you felt downhearted and depressed? (Variable(s): W102_RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, column and row totals, ynominal proportion (if any). | | ` ′ | | X |
| Have you felt downhearted and depressed? (Variable(s): MH04 RESPONSE) Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal Qualitative, nominal Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, x | (variable(s): v102_KESPONSE) | nominai | | |
| depressed? Qualitative, nominal column and row totals, missing proportion (if any). X Did you feel worn out? Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). X Have you been happy? Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, column and row totals, X | Have you felt downhearted and | Oval!4-4!- | | |
| (Variable(s): MH04 RESPONSE) nominal missing proportion (if any). Did you feel worn out? (Variable(s): VT03_RESPONSE) Qualitative, nominal missing proportions, frequencies, column and row totals, missing proportion (if any). Have you been happy? (Variable(s): MH05_RESPONSE) Qualitative, propringly proportions, frequencies, column and row totals, | | 1 ' | | X |
| Did you feel worn out? Qualitative, nominal Proportions, frequencies, column and row totals, missing proportion (if any). X Have you been happy? Qualitative, propringly column and row totals, nominal Proportions, frequencies, column and row totals, column and row totals, X | | nominai | | |
| (Variable(s): VT03_RESPONSE) Qualitative, nominal column and row totals, missing proportion (if any). Proportions, frequencies, column and row totals, (Variable(s): MH05_RESPONSE) Qualitative, rominal row totals, missing proportion (if any). | | O1'(-1' | | |
| (Variable(s): V103_RESPONSE) nominal missing proportion (if any). Proportions, frequencies, column and row totals, X | | 1 ' | | X |
| Have you been happy? (Variable(s): MH05_RESPONSE) Qualitative, column and row totals, X | (variable(s): v103_RESPONSE) | nominal | | |
| (Variable(s): MH05 RESPONSE) Qualitative, column and row totals, | Harraman has the exp | O1'(1' | | |
| | | | | X |
| | (variable(s): MHU3_KESPONSE) | nominai | | |

| | 1 | D | 1 | 1 | 1 |
|---|---|---|---|---|---|
| Did you feel tired? | Qualitative, | Proportions, frequencies, column and row totals, | | | X |
| (Variable(s): VT04_RESPONSE) | nominal | missing proportion (if any). | | | |
| During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting friends, relatives, etc.)? (Variable(s): SF02 RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| I seem to get sick a little easier than | | Proportions, frequencies, | | | |
| other people (Variable(s): GH02_RESPONSE) | Qualitative, nominal | column and row totals, missing proportion (if any). | | | X |
| I am as healthy as anybody I know<br>(Variable(s): GH03_RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| I expect my health to get worse<br>(Variable(s): GH04_RESPONSE) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| My health is excellent (Variable(s): GH05_RESPONSE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Physical Functioning<br>(Variable(s): PFSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Role Physical<br>(Variable(s): RPSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | х | X | |
| Bodily Pain<br>(Variable(s): BPSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| General Health<br>(Variable(s): GHSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Vitality<br>(Variable(s): VTSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, | X | X | |

| | | . 1 11 1 050/ | | | 1 |
|---|---|---|---|---|---|
| | | standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | |
| Social Functioning<br>(Variable(s): SFSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Role Emotional<br>(Variable(s): RESCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | х | |
| Mental Health<br>(Variable(s): MHSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Total Physical Score<br>(Variable(s): PCSSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | Х | |
| Total Mental Score<br>(Variable(s): MCSSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | X | |

Table 6.5.2: Post-Operative Visit Form – SF-36 Score Tables List

### 6.6. ANALYSIS OF CI ENDPOINTS

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan |
|-----------------------------------|-------------------------|---------------|
| Fuducints - Primary Fuducint | | |

#### Endpoints – Primary Endpoint

Use variable SF-36 Total Physical Score 12 Months [points]:

Based on the underlying distribution of the data and the result of the normality assessment, either the parametric one-sample t-test or the non-parametric one-sample sign test will be used to compare the 12 months post-operative SF-36 score results of the T2 Alpha Tibia group against the value of 39.25 points.

The complete available SPSS tables content related to either the one-sample t-test or the one-sample sign test will be included in the <u>final report</u> (under no circumstances, creation of this analysis in any interim/annual report). (Variable(s): VISITDT; PCSSCORE)

Table 6.6.1: Endpoints – Primary Endpoint Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recode and Analysis<br>Plan | Ir | ıclusio | n |
|---|---|---|---|---|---|
| All Assessments – Fracture Healing | | | IR | FR | N/A |
| 3 Months - 4. Has the bone consolidated (consider weightbearing, pain and imaging)? (Variable(s): VISITDT; BONECONS) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| 6 Months - 4. Has the bone consolidated (consider weight-bearing, pain and imaging)? (Variable(s): VISITDT; BONECONS) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| 12 Months - 4. Has the bone consolidated (consider weight-bearing, pain and imaging)? (Variable(s): VISITDT; BONECONS) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |

Table 6.6.2: Endpoints – Secondary Endpoint Fracture Healing Tables List

| Evaluation | Level of | Recode and Analysis | т | , . | |
|---|---|---|---|---|---|
| Variable / Question | Measurement | Ir | ıclusio | n | |
| Adverse Events – Time to (earliest) Device Related Adverse Event/ | | | | | N/A |
| Incident | | | | FR | IN/A |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of First Device Related Adverse Event [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT; VISNAME; AEONSTDT) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of 12 Months Visit [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT; VISNAME) | Quantitative,<br>ratio | N/A (Analyzed above), used for survivorship | | X | |
| Create new variable "Grouping variable – First Device Related Adverse Event" (Variable(s): AEEVENT) | Qualitative,<br>nominal | - censored = survivors<br>- events = first (earliest) Device<br>Related Adverse Event | | Х | |
| Create new variable "Combined Time – First Device Related Adverse Event" (Variable(s): AEONSTDT) | Quantitative, ratio | Use time between surgery and 12 months visit for surviving subjects Use time between surgery and first device related adverse event for subjects with device related adverse event | | X | |
| Use variables "Combined Time – First<br>Device Related Adverse Event" | Qualitative, | Case summary with number and percentage of valid | | X | |

| and "Grouping variable - First Device | nominal | cases/values, missing |
|---|---|---|
| Related Adverse Event" | Quantitative, | cases/values (if any) and total |
| | ratio | cases/values. |
| | | Kaplan-Meier survival |
| | | analysis: subject ID, time, |
| | | status, cumulative proportion, |
| | | Kaplan-Meier estimate, |
| | | standard error of KM estimate, |
| | | number of cumulative events, |
| | | number of remaining cases, |
| | | mean for survival time with |
| | | 95% confidence interval, |
| | | survival graph, hazard graph. |

Table 6.6.3: Endpoints – Secondary Endpoint Time to (earliest) Device Related Adverse Event / Incident Tables List

### 6.7. ADDITIONAL ANALYSIS

### 6.7.1.SF-36 Total Physical Score Comparison

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan |
|---|---|---|
|---|---|---|

### All Assessments – SF-36 Total Physical Score Comparison

Use "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 3 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 3 Months [points]" to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Use "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 6 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 6 Months [points]" to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Use "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 12 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total Physical Score Pre-Op [points]" and "SF-36 Total Physical Score 12 Months [points]" to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Use "SF-36 Total Physical Score 3 Months [points]" and "SF-36 Total Physical Score 6 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total Physical Score 3 Months [points]" and "SF-36 Total Physical Score 6 Months [points]": to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Use "SF-36 Total Physical Score 3 Months [points]" and "SF-36 Total Physical Score 12 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total Physical Score 3 Months [points]" and "SF-36 Total Physical Score 12 Months [points]": to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Use "SF-36 Total Physical Score 6 Months [points]" and "SF-36 Total Physical Score 12 Months [points]": Based on the underlying distribution of the data in both groups and the result of the normality assessment, either the parametric paired samples t-test or the non-parametric Wilcoxon test will be used to compare "SF-36 Total

*Physical Score 6 Months [points]"* and "SF-36 Total Physical Score 12 Months [points]": to evaluate the SF-36 PCS score change by subject (improvement or decrease).

The complete available SPSS tables content related to either the paired samples t-test or the Wilcoxon test will be included in the final report.

(Variable(s): VISITDT; PCSSCORE)

Table 6.7.1: All Assessments – SF-36 Total Physical Score Comparison Tables List

### 6.7.2. Weight-bearing status

As listed above, the weight bearing status will be evaluated and analyzed at the preoperative visit and at 3 months, 6 months and 12 months. The within subject changes from visit to visit will be analyzed in addition. This analysis is part of the final report.

The variable capturing weight bearing will be used with "yes" (including partial and full) versus "no" weightbearing.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recoding |
|---|---|---|
| All Assessments - Weight-b | | |
| Recode initial weightbearing status at pre-op visit into new variable "Pre-Op Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative, nominal | The initial variable capturing weight bearing preop will be recoded with "yes" (including partial and full) versus "no" weightbearing. |
| Recode initial weightbearing status at pre-op visit into new variable "3 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | The initial variable capturing weight bearing at 3 months will be recoded with "yes" (including partial and full) versus "no" weightbearing. |
| Recode initial weightbearing status at pre-op visit into new variable "6 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | The initial variable capturing weight bearing at 6 months will be recoded with "yes" (including partial and full) versus "no" weightbearing. |
| Recode initial weightbearing status at pre-op visit into new variable "12 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | The initial variable capturing weight bearing at 12 months will be recoded with "yes" (including partial and full) versus "no" weightbearing. |

Table 6.7.2.1: All Assessments – Weight-bearing status Recoding

New variables (10) will then be created for each possible pair/comparison. Negative changes (from "yes" to "no") will be coded with "negative change" and positive changes (from "no" to "yes") with be coded with "positive change". If there is no change (from "yes" to "yes" or from "no" to "no"), the coding will be "no change".

| Evaluation<br>Variable / Question | Level of<br>Measurement | Coding and Analysis Plan |
|---|---|---|
| All Assessments - Weight-bearing state | us | |
| Create new variable "Weightbearing status change between pre-operative visit and 3 months" based on comparison of "Pre-Op Weightbearing Dichotomous" with "3 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and row totals, missing proportion (if any). |

| Create new variable "Weightbearing status change between pre-operative visit and 6 months" based on comparison of "Pre-Op Weightbearing Dichotomous" with "6 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and row totals, missing proportion (if any). |
|---|---|---|
| Create new variable "Weightbearing status change between pre-operative visit and 12 months" based on comparison of "Pre-Op Weightbearing Dichotomous" with "12 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and |
| Create new variable "Weightbearing status change between 3 months and 6 months" based on comparison of "3 Months Weightbearing Dichotomous" with "6 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | row totals, missing proportion (if any). - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and |
| Create new variable "Weightbearing status change between 3 months and 12 months" based on comparison of "3 Months Weightbearing Dichotomous" with "12 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | row totals, missing proportion (if any). - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and row totals, missing proportion (if any). |
| Create new variable "Weightbearing status change between 6 months and 12 months" based on comparison of "6 Months Weightbearing Dichotomous" with "12 Months Weightbearing Dichotomous" (Variable(s): VISITDT; WEIGHTBEAR) | Qualitative,<br>nominal | - Negative changes (from "yes" to "no") = "negative change" - Positive changes (from "no" to "yes") = "positive change" - No change (from "yes" to "yes" or from "no" to "no") = "no change" Proportions, frequencies, column and row totals, missing proportion (if any). |

Table 6.7.2.2: All Assessments – Weight-bearing status Tables List

### 6.7.3. External Support

As listed above, the status of the subject using external support will be evaluated at the preoperative visit and at 3 months, 6 months and 12 months. The within subject changes from visit to visit will be analyzed in addition. This analysis is part of the final report.

The variable capturing "Is the subject using an external support" will be used and recoded into a new variable for each visit with the options "no" (using no support at all) versus "yes" (including Walker, Cane, One Crutch or Two Crutches).

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recoding |
|---|---|---|
| All Assessments – Extern | al support stat | us |
| Recode initial external support status at pre-op visit into new variable "Pre-Op External Support Dichotomous" (Variable(s): EXTRSUPP) | Qualitative,<br>nominal | The variable capturing "Is the subject using an external support" will be used and recoded into a new variable for each visit with the options "no" (using no support at all) versus "yes" (including Walker, Cane, One Crutch or Two Crutches). |
| Recode initial external support status at pre-op visit into new variable "3 | Qualitative,<br>nominal | The variable capturing "Is the subject using an external support" will be used and recoded into a new variable for each visit with the options "no" (using no support at all) |

| Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | | versus "yes" (including Walker, Cane, One Crutch or Two Crutches). |
|---|---|---|
| Recode initial external support<br>status at pre-op visit into new<br>variable "6 Months External<br>Support Dichotomous"<br>(Variable(s): VISITDT;<br>EXTRSUPP) | Qualitative,<br>nominal | The variable capturing "Is the subject using an external support" will be used and recoded into a new variable for each visit with the options "no" (using no support at all) versus "yes" (including Walker, Cane, One Crutch or Two Crutches). |
| Recode initial external support<br>status at pre-op visit into new<br>variable "12 Months External<br>Support Dichotomous"<br>(Variable(s): VISITDT;<br>EXTRSUPP) | | The variable capturing "Is the subject using an external support" will be used and recoded into a new variable for each visit with the options "no" (using no support at all) versus "yes" (including Walker, Cane, One Crutch or Two Crutches). |

Table 6.7.3.1: All Assessments – External Support Recoding

New variables (10) will then be created for each comparison listed below. Negative changes (from "no" to "yes") will be coded with "negative change" and positive changes (from "yes" to "no") with be coded with "positive change". If there is no change (from "yes" to "yes" or from "no" to "no"), the coding will be "no change".

| Evaluation<br>Variable / Question | Level of<br>Measurement | Coding and Analysis Plan |
|---|---|---|
| All Assessments - External support status | | |
| Create new variable "External support status change between preoperative visit and 3 months" based on comparison of "Pre-Op External Support Dichotomous" with "3 Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> <li>Proportions, frequencies, column and row totals, missing proportion (if any).</li> </ul> |
| Create new variable "External support status change between pre- operative visit and 6 months" based on comparison of "Pre-Op External Support Dichotomous" with "6 Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> <li>Proportions, frequencies, column and row totals, missing proportion (if any).</li> </ul> |
| Create new variable "External support status change between pre- operative visit and 12 months" based on comparison of "Pre-Op External Support Dichotomous" with "12 Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> <li>Proportions, frequencies, column and row totals, missing proportion (if any).</li> </ul> |
| Create new variable "External support status change between 3 months and 6 months" based on comparison of "3 Months External Support Dichotomous" with "6 | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> </ul> |

| Months External Support<br>Dichotomous"<br>(Variable(s): VISITDT;<br>EXTRSUPP) | | Proportions, frequencies, column and row totals, missing proportion (if any). |
|---|---|---|
| Create new variable "External support status change between 3 months and 12 months" based on comparison of "3 Months External Support Dichotomous" with "12 Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> <li>Proportions, frequencies, column and row totals, missing proportion (if any).</li> </ul> |
| Create new variable "External support status change between 6 months and 12 months" based on comparison of "6 Months External Support Dichotomous" with "12 Months External Support Dichotomous" (Variable(s): VISITDT; EXTRSUPP) | Qualitative,<br>nominal | <ul> <li>Negative changes (from "yes" to "no") = "negative change"</li> <li>Positive changes (from "no" to "yes") = "positive change"</li> <li>No change (from "yes" to "yes" or from "no" to "no") = "no change"</li> <li>Proportions, frequencies, column and row totals, missing proportion (if any).</li> </ul> |

Table 6.7.3.2: All Assessments – External support status Tables List

### 6.7.4. Mortality

For analysis of the time to death or mortality, the Kaplan-Meier method will be used. The times between surgery and the 12 months assessment will be used together with the times between surgery and the date of death. This analysis is part of the final report.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recode and Analysis Plan |
|---|---|---|
| All Assessments - Morta | All Assessments - Mortality | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of Death [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT; DOSEDD) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of 12 Months Visit [dd.mm.yyyy] in days J (Variable(s): VISITDT) | Quantitative, ratio | N/A (Analyzed above), used for survivorship |
| Create new variable "Grouping variable - Mortality" (Variable(s): PRIMRSN) | Qualitative,<br>nominal | - censored = survivors<br>- events = death |
| Create new variable "Combined Time - Mortality" (Variable(s): VISITDT; DOSEDD) | Quantitative, ratio | Use time between surgery and 12 months visit for surviving subjects Use time between surgery and death for deceased subject |

| Use variables "Combined<br>Time -<br>Mortality" and "Grouping<br>variable - Mortality" | Qualitative,<br>nominal<br>Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Kaplan-Meier survival analysis: subject ID, time, status, cumulative proportion, Kaplan-Meier estimate, standard error of KM estimate, number of cumulative events, number of remaining cases, mean for survival time with 95% confidence interval, survival graph, hazard graph. |
|---|---|---|
|---|---|---|

Table 6.7.4: All Assessments – Mortality Tables List

### 6.7.5. Revision Surgery

For analysis of the time to the revision surgery, the Kaplan-Meier method will be used. The times between surgery and the 12 months assessment will be used together with the times between surgery and the date of revision (earliest revision in case that one subject experienced more than one revision). This analysis is part of the final report.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recode and Analysis Plan |
|---|---|---|
| Adverse Events / Revision Surgery | | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of First Revision [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of 12 Months Visit [dd.mm.yyyy] in days (Variable(s): VISITDT) | Quantitative, ratio | N/A (Analyzed above), used for survivorship |
| Create new variable "Grouping variable – First Revision" (Variable(s): VISITDT) | Qualitative,<br>nominal | - censored = survivors<br>- events = first (earliest) Revision |
| Create new variable "Combined Time – First Revision" (Variable(s): VISITDT) | Quantitative, ratio | <ul> <li>Use time between surgery and 12 months visit for surviving subjects</li> <li>Use time between surgery and first revision for subjects with revision(s)</li> </ul> |
| Use variables "Combined<br>Time – First<br>Revision" and "Grouping<br>variable – First Revision" | Qualitative,<br>nominal<br>Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Kaplan-Meier survival analysis: subject ID, time, status, cumulative proportion, Kaplan-Meier estimate, standard error of KM estimate, number of cumulative events, number of remaining cases, mean for survival time with 95% confidence interval, survival graph, hazard graph. |

Table 6.7.5: All Assessments – Revision Surgery Tables List

### 6.7.6. SF-36 Total Physical Score – Within subject changes by visit

The within subject score changes of the SF-36 Total Physical Score from visit to visit will be analyzed to help identifying the changes on the subject level. This analysis is part of the report.

| | Measurement | Coding and Analysis Plan in Subject Changes |
|---|---|---|
| Creation of variable "SF-36 Total Physical Score change between pre-operative visit and 3 Months [points]" | Quantitative, interval | Calculate difference (could be negative or positive). |

| D:# 1 . #GE 26 T. (1D) * 1 | | 0 21 1 1 |
|---|---|---|
| Difference between "SF-36 Total Physical Score Pre-Op [points]" with "SF-36 Total Physical Score 3 Months [points]" (Variable(s): VISITDT; PCSSCORE) | | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable "SF-36 Total Physical Score change between pre-operative visit and 6 Months [points]" Difference between "SF-36 Total Physical Score Pre-Op [points]" with "SF-36 Total Physical Score 6 Months [points]" (Variable(s): VISITDT; PCSSCORE) | Quantitative, interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable "SF-36 Total Physical Score change between pre-operative visit and 12 Months [points]" Difference between "SF-36 Total Physical Score Pre-Op [points]" with "SF-36 Total Physical Score 12 Months [points]" (Variable(s): VISITDT; PCSSCORE) | Quantitative, interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable "SF-36 Total Physical Score change between 3 Months and 6 Months [points]" Difference between "SF-36 Total Physical Score 3 Months [points]" with "SF-36 Total Physical Score 6 Months [points]" (Variable(s): VISITDT; PCSSCORE) | Quantitative, interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable "SF-36 Total Physical Score change between 3 Months and 12 Months [points]" Difference between "SF-36 Total Physical Score 3 Months [points]" with "SF-36 Total Physical Score 12 Months [points]" (Variable(s): VISITDT; PCSSCORE) | Quantitative,<br>interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable "SF-36 Total Physical<br>Score change between 6 Months and 12<br>Months [points]"<br>Difference between "SF-36 Total Physical<br>Score 6 Months [points]" with "SF-36 Total<br>Physical Score 12 Months [points]"<br>(Variable(s): VISITDT; PCSSCORE) | Quantitative, interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |

Table 6.7.6: All Assessments – SF-36 Total Physical Score Within Subject Changes

### 7. Table Templates (Tables, Figures, Listings - TFL)

Tables must consist of at least a headline, the variable/analysis-object label and column headers. Furthermore, the table headline must contain the "Analysis Section" (e.g. Demographics, Operative) the variable label (e.g. Gender, Age) as well as the table type (Frequencies, Listing). If the table is referring to a subgroup, a notification must be entered in the headline as well. Figures (if any) must be clearly labeled and numbered by a figure number and title in addition to the axis and category labeling created by software packages (e.g. IBM SPSS).

### 7.1. FREQUENCIES

All answered response options must be listed with the appropriate label, other response options do not have to be displayed necessarily. In the event of missing answers, the frequencies must be included in an extra row as well ("Missing"). All given answers must be added up in an extra row ("Total"). In addition to the number of frequencies, percentages must be displayed in a separate column.

| "Analysis Section" | " – "Variable | Label" - | <b>Frequencies</b> |
|------------------------|---------------|----------|-----------------------|
| 1 Illiery StS & Cetton | , | | I . Cy W. C. W. C. C. |

| Characteristic | | n | % |
|------------------|--------------|-------|-------|
| | "Response A" | "xxx" | "xxx" |
| "Variable Label" | "Response B" | "xxx" | "xxx" |
| v ariabie Labei | Missing | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" |

Table 7.1.1: Frequencies Table Template

If multiple subgroups/clusters (e.g. Sites, Visits) should be displayed in one table, an extra column ("Group X") and/or extra rows ("Group Y") must be added. Same applies to (sub-) questions, which can be merged in one table. It is recommended to add an extra "Total" column and row, for adding up the subgroups, if possible, from a statistical point of view. In addition, subgroups must be named in the headline as well ("by Group X and by Group Y").

"Analysis Section" – "Variable Label" – Frequencies – by "Group X" and "Group Y"

| Group 1 | | | | | | | |
|---|---|---|---|---|---|---|---|
| Chanastanisti | Characteristic | | "Group X1" | | "Group X2" | | Total |
| Characteristi | | | % | n | % | n | % |
| | "Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Crown VI" | "Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Group Y1" | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | "Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Crown V2 | "Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Group Y2 | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | "Total Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| T-4-1 | "Total Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| Total | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |

Table 7.1.2: Grouped Frequencies Table Template

### 7.2. DESCRIPTIVE STATISTICS

Descriptive Statistic tables must contain the items listed in Table 7.2.1. Furthermore, the associated unit must be displayed. If the values are referring to a subgroup (n) and not to the overall population (N), a notification must be entered in the headline ("n = xxx").

### "Analysis Section" – "Variable Label" – Descriptive Statistics (n = "xxx")

| Characteristic | | ["unit"] |
|------------------|--------|----------|
| | Mean | "xxx" |
| | Median | "xxx" |
| "I/:l.1 - Il1" | SD | "xxx" |
| "Variable Label" | IQR | "xxx" |
| | Max | "xxx" |
| | Min | "xxx" |

Table 7.2.1: Descriptive Statistics Table Template

### 7.3. LISTINGS

Listing tables must contain one unique identifier (e.g. Subject ID). Furthermore, an additional column must be added, if the specification/description is not referring to one single variable or response option("Response Option"), which is already named in the headline. If multiple specifications/descriptions exist for one variable/response (e.g. Drug1, Drug2, Drug3...), further columns must be added ("Specification/Description A", "Specification/Description B"). Subgroups can be implemented as described in chapter 7.1.

### "Analysis Section" - "Variable Label" - Listing

| "Unique | Description | |
|-------------|-------------------|-------------------------------|
| Identifier" | "Response Option" | "Specification/Description A" |
| "xxx" | "xxx" | "xxx" |
| "xxx" | "xxx" | "xxx" |
| "xxx" | "xxx" | "xxx" |

Table 7.3.1: Listing Table Template

### 8. References

- a. ISO 14155 Clinical Investigation of Medical Devices for Human Subjects
- b. ICH-E6 Harmonized Tripartite Guidelines for Good Clinical Practice
- c. ICH-E9 Statistical Principles for Clinical Trials
- d. Declaration of Helsinki
- e. Gamble C et. al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. AMA. 2017;318(23):2337-2343. doi:10.1001/jama.2017.18556
- f. DQP 20-001 Clinical Investigation
- g. DQI 20-001 Clinical Investigation Clinical Investigation Plan
- h. DQI 20-004 Clinical Investigation Master CRF, eCRF and Database Development
- i. DQI 20-009 Clinical Investigation Reports

# 20210723\_T2 Alpha Tibia\_SAP

Final Audit Report 2021-07-23

Created: 2021-07-23

By: Sascha Lorenzen (sascha.lorenzen@stryker.com)

Status: Signed

Transaction ID: CBJCHBCAABAAi2TVOC2kT-sjeSuSIVbO8abj4xnwxP40

# "20210723\_T2 Alpha Tibia\_SAP" History

- Document created by Sascha Lorenzen (sascha.lorenzen@stryker.com) 2021-07-23 10:12:37 AM GMT- IP address: 89.15.237.222
- Document emailed to Sascha Lorenzen (sascha.lorenzen@stryker.com) for signature 2021-07-23 10:14:22 AM GMT
- Document emailed to Claudia Beimel (claudia.beimel@stryker.com) for signature 2021-07-23 10:14:22 AM GMT
- Document emailed to Rebecca Gibson (rebecca.gibson@stryker.com) for signature 2021-07-23 10:14:22 AM GMT
- Document emailed to Susanne Höfer (susanne.hoefer@stryker.com) for signature 2021-07-23 10:14:22 AM GMT
- Sascha Lorenzen (sascha.lorenzen@stryker.com) verified identity with Adobe Sign authentication 2021-07-23 - 10:15:53 AM GMT
- Document e-signed by Sascha Lorenzen (sascha.lorenzen@stryker.com)

  Signature Date: 2021-07-23 10:15:53 AM GMT Time Source: server- IP address: 89.15.237.222
- Email viewed by Susanne Höfer (susanne.hoefer@stryker.com) 2021-07-23 10:34:07 AM GMT- IP address: 87.169.18.160
- Susanne Höfer (susanne.hoefer@stryker.com) verified identity with Adobe Sign authentication 2021-07-23 10:36:23 AM GMT
- Document e-signed by Susanne Höfer (susanne.hoefer@stryker.com)
  Signature Date: 2021-07-23 10:36:23 AM GMT Time Source: server- IP address: 87.169.18.160
- Claudia Beimel (claudia.beimel@stryker.com) verified identity with Adobe Sign authentication 2021-07-23 - 11:19:01 AM GMT



- Document e-signed by Claudia Beimel (claudia.beimel@stryker.com)

  Signature Date: 2021-07-23 11:19:01 AM GMT Time Source: server- IP address: 195.243.167.66
- Email viewed by Rebecca Gibson (rebecca.gibson@stryker.com) 2021-07-23 4:23:20 PM GMT- IP address: 52.154.71.15
- Rebecca Gibson (rebecca.gibson@stryker.com) verified identity with Adobe Sign authentication 2021-07-23 4:35:51 PM GMT
- Document e-signed by Rebecca Gibson (rebecca.gibson@stryker.com)

  Signature Date: 2021-07-23 4:35:51 PM GMT Time Source: server- IP address: 52.154.71.15
- Agreement completed.
   2021-07-23 4:35:51 PM GMT